CLINICAL TRIAL: NCT04754620
Title: Implementation and Evaluation of Smartphone-Based Videoconferance Telehealth for Patients With Crohn's Disease
Brief Title: Distant Management of Crohn's Disease by Smartphones is Feasible and Effective Additionally it Reduces the Costs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hasan Yılmaz, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KouTeleH001
Record Dates: First submitted 2021-02-05; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard face to face visit (No Intervention): This group will receive a traditional outpatient visit
- Online visit (Experimental): This group will receive a smartphone-based real-time video conference visit
  Interventions: Other: real time online video visit

INTERVENTIONS:
Other: real time online video visit — Participants have received an online visit by a smartphone application
  Arms: Online visit

SUMMARY:
Evaluation of the feasibility, acceptability, patient satisfaction and economic benefits of smartphone video-based telehealth in the management of Crohn's disease patients

DETAILED DESCRIPTION:
Patients were examined by two gastroenterologists (HY, AED) either at a video conference based visit or face to face visit in outpatients clinics. We used the WhatsApp business application.The online visit notion was the same as traditional face-to-face visit except physical examination.

ELIGIBILITY:
Inclusion Criteria:

* The study group included patients with documented Crohn's disease, based on clinical, endoscopic, and histologic findings
* Patient between 18-80 years old
* Participants who have been receiving treatment for more than six months

Exclusion Criteria:

* Patients were excluded from the study if they had no internet connection
* Unable to use smartphones because of blindness, deafness, or mental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction score with the video visits | the day after the visit
  Measurement of satisfaction with RAND Visit Specific Questionnaire (VSQ9),Minimum score "0" poor and maximum score is "5" represents excellent,

CONTACTS AND LOCATIONS:
Overall Officials: göktuğ şirin, Study Director — Kocaeli University
Locations (1):
- Kocaeli University Medical Faculty Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code
Time Frame: Data will be available for one year after the study completed
Access Criteria: Public